CLINICAL TRIAL: NCT04548973
Title: A Multicenter Study of the Efficacy and Safety of Esketamine for Analgesia During
Brief Title: A Multicenter Study of the Efficacy and Safety of Esketamine for Analgesia During Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MZK20200831
Record Dates: First submitted 2020-08-31; First posted 2020-09-16 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Fetal or Neonatal Effect of Damage to Placenta From Caesarean Section
Keywords: Esketamine, cesarean section, parturient, placental transfer
MeSH Terms: interventions — Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine Group (Experimental): At the beginning of the operation, 0.25mg/kg ketamine was administered intravenously, and normal saline was diluted to 2mL to assist sedation and analgesia
  Interventions: Drug: Esketamine
- Control Group (Placebo Comparator): At the beginning of the operation, 2ml normal saline was given intravenously
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Esketamine — Esketamine
  Arms: Esketamine Group
Drug: Normal saline — 2ml normal saline
  Arms: Control Group

SUMMARY:
This study proposed applying intravenous Esketamine to cesarean section in parturient, detecting the plasma concentration of Esketamine in maternal blood, neonatal umbilical venous blood and umbilical arterial blood when the baby is delivered ketamine blood drug concentration, observing vital signs, adverse visual analog pain score (VAS), and sedation score (Ramsay) in parturient, neonatal Apgar score 1, 5 to 10 minutes after birth, the umbilical arterial blood gas and neurobehavioral scores (NBNA) 2, 24 hours after the birth. This study aims to address placental transfer, metabolism and analgesic and sedative effects in neonates and parturients of Esketamine so as to explore the feasibility, efficacy and safety of Esketamine as adjuvant medication for cesarean section.

DETAILED DESCRIPTION:
1. case selection: A total of 600 patients (American Society of Anesthesiologists (ASA) grade I-II, aged 20-40 years,BMI 18.5-27) who underwent elective cesarean section were selected.
2. anesthesia methods: All patients were not given preoperative medication. After entering the operating room, peripheral venous connection was opened. Mindray multifunctional vital sign monitor continuously monitored electrocardiogram (ECG), heart rate (HR), pulse oxygen saturation (SpO2), systolic blood pressure (SBP), diastolic blood pressure (DBP) and Mean arterial pressure (MAP). After 5 minutes of waiting for patients with no obvious discomfort, 0.75% of ropivacaine was given 10ml before catheterization, and 0.75% of ropivacaine 3-5ml per hour maintained anesthesia
3. Grouping methods: A random number table was used to divide the patients into two groups with 300 patients in each group: The Esketamine group (group A) and the control group (group B) Esketamine group (Group A): at the beginning of the operation, 0.25mg/kg(2ml) Esketamine was administered intravenously as an adjuvant sedation and analgesia;Control group (Group B): 2ml normal saline was given intravenously at the beginning of the operation;
4. Observation items and methods 4.1 Forty patients were randomly selected from the Estroketamine group (group A) to detect the serum concentrations of Esketamine in umbilical vein blood and umbilical artery blood of neonates during fetal delivery.

4.2 maternal hemodynamic indexes such as heart rate (HR), mean arterial pressure (MAP) and respiratory mechanics indexes such as pulse oxygen saturation (SpO2) and shout at the end of the co2 partial pressure (PaCO2) are measured before anesthesia surgery at the beginning of the fetal childbirth at the end of the operation and operation after 1 hour when recording and compare the two groups of 4.3 maternal visual analog pain score (VAS) and sedation scores (Ramsay) and the time from uterine incision to fetal childbirth are measured before anesthesia surgery at the beginning of the fetal childbirthAt the end of the operation and operation after 1 hour record and compare the two groups of 4.4 respiratory system complications within 72 h in pregnant women (hypotension sinus bradycardia nausea and vomiting respiratory depression) are record.

4.5 Apgar score 1, 5, 10 minutes after birth, umbilical arterial blood gas and neurobehavioral scores (NBNA) 2 and 24 hours after the birth are record.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* full-term single pregnancy
* had regular prenatal examination
* scheduled for elective cesarean delivery with epidural anesthesia

Exclusion Criteria:

* body mass index (calculated as weight in kilograms divided by height in meters squared) of 27 or greater
* previous mental illness, central nervous system disease, liver disease, abnormal kidney function, abnormal heart and lung function, diabetes, or American Society of Anesthesiologists (ASA) classification III or above
* severe obstetric complications, such as preeclampsia and eclampsia, pregnancy-induced hypertension, placenta previa, or placental abruption
* stillbirth or neonatal malformation
* contraindications to epidural anesthesia, including abnormal coagulation function, anticoagulant therapy, severe hypovolemia, or hemodynamic instability

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — parturient
Enrollment: 600 (Actual)
Dates: Start 2021-09-18 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Maternal pain intensity | immediately after fetal delivery
  Pain intensity was assessed with the numeric rating scale (NRS; an 11-point scale, with 0 indicating no pain and 10 indicating the worst pain)
Maternal sedation level | immediately after fetal delivery
  Maternal sedation level was assessed with Ramsay Sedation Scale (with 1 indicating restless; 2, completely awake, quiet, and cooperative; 3, drowsy but responding to verbal commands; 4, lightly asleep but responding to touch or pain; 5, asleep but slowly responding to touch or pain; and 6, deeply asleep and does not respond)

SECONDARY OUTCOMES:
Maternal pain intensity at other timepoints | before anesthesia, immediately after anesthesia, surgical incision, 5 minutes after study, end of surgery, 6 hours after surgery, and 12 hours after surgery. drug administration,
  Maternal pain intensity at other timepoints were assessed with the numeric rating scale (NRS; an 11-point scale, with 0 indicating no pain and 10 indicating the worst pain)
Maternal sedation level at other timepoints | before anesthesia, immediately after anesthesia, surgical incision, 5 minutes after study, end of surgery, 6 hours after surgery, and 12 hours after surgery. drug administration,
  Maternal sedation level at other timepoints were assessed with Ramsay Sedation Scale (with 1 indicating restless; 2, completely awake, quiet, and cooperative; 3, drowsy but responding to verbal commands; 4, lightly asleep but responding to touch or pain; 5, asleep but slowly responding to touch or pain; and 6, deeply asleep and does not respond)
systolic blood pressure, diastolic blood pressure, and mean blood pressure | before anesthesia, immediately after anesthesia, at surgical incision, 5 minutes after study drug administration, immediately after fetal delivery, at end of surgery, and 1 hour after surgery
  systolic and diastolic blood pressure were assessed by non-invasive blood pressure cuff，mean blood pressure was measured by the Calculation formula: Mean arterial pressure =(systolic pressure +2× diastolic pressure)/3
maternal heart rate | before anesthesia, immediately after anesthesia, at surgical incision, 5 minutes after study drug administration, immediately after fetal delivery, at end of surgery, and 1 hour after surgery
  maternal heart rate
pulse oxygen saturation | before anesthesia, immediately after anesthesia, at surgical incision, 5 minutes after study drug administration, immediately after fetal delivery, at end of surgery, and 1 hour after surgery
  pulse oxygen saturation
Apgar score of newborn | at 1 minute and 5 minute after birth
  Apgar was assessed by appearance, pulse, grimace, activity, respiration. Each item was measured on a scale of 0, 1, and 2, respectively, with a maximum total score of 10.
postnatal umbilical vein blood gas pH value | Results of umbilical arterial blood gas analysis after birth
  postnatal umbilical vein blood gas pH value
Esketamine concentrations in maternal arterial blood and neonatal umbilical arterial | Immediately after fetal delivery
  Esketamine concentrations was assessed by reverse-phase high-performance liquid chromatography

OTHER OUTCOMES:
Adverse events including hypotension, hypertension, bradycardia, tachycardia and desaturation | Adverse events were recorded as Frequency of occurrence between the time the patient entered the operating room and the end of surgery
  hypotension was defined as a systolic blood pressure decrease less than 20% of baseline, hypertension was defined as a systolic blood pressure increase greater than 20% of baseline, bradycardia was defined as a heart rate less than 60 beats per minute, tachycardia was defined as a heart rate greater than 100 beats per minute, and desaturation was defined as oxygen saturation less than 90%.
offspring's neurodevelopment | 2 years after birth
  Neurodevelopment was measured by the Ages and Stages Questionnaire, third edition (ASQ-3).The ASQ-3 assesses 5 developmental domains: gross motor skills, fine motor skills, problem-solving ability, communication, and personal and social skills. Each domain is assessed by 6 questions ascertaining achievement of relevant skills and answered as yes (10 points), sometimes (5 points), or not yet (0 points). Scores for individual items are summed to give an overall continuous score for each of the 5 domains (possible range, 0-60).
Mothers' memories of childbirth | at 2 years after birth
  Mothers' memories of childbirth was assessed by The Birth Memories and Recall Questionnaire (BirthMARQ),which focused on parents' positive, negative or mixed emotions at the birth/in recalling the event. Each item (e.g. 'my emotions at the time were extremely negative') was rated on a scale ranging from 1 (strongly disagree) to 7 (strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu LL, Wang C, Deng CM, Dai SB, Zhou Q, Peng YB, Shou HY, Han YQ, Yu J, Liu CH, Xia F, Zhang SQ, Wang DX, Chen XZ. Efficacy and Safety of Esketamine for Supplemental Analgesia During Elective Cesarean Delivery: A Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e239321. doi: 10.1001/jamanetworkopen.2023.9321. PMID 37083664

DOCUMENTS (1):
  • Study Protocol (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/73/NCT04548973/Prot_000.pdf